CLINICAL TRIAL: NCT02429206
Title: Prospective, Double Blind, Randomized Phase II/III Study to Assess the Safety and Efficacy of SQIN™ on Xerosis in Adults Suffering of Mobility Impairment and/or Complete Paralysis Associated With Chronic Spinal Cord Injury.
Brief Title: Safety and Efficacy of SQIN™ on Xerosis in Adults With Mobility Problems and Paralysis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nordic Life Science Pipeline Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SQIN-01
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Xerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Control (Active Comparator): Each volunteer will be asked to self-apply a standard moisturizing cream (Glaxal Base) on one side of their body. Application twice a day during 14 days.
  Interventions: Other: standard moisturizing cream (Glaxal Base)
- Experimental Cream (Experimental): Each volunteer will be asked to self-apply the experimental product (SQIN with CanSATs technology) on the other side of their body. Application twice a day during 14 days.
  Interventions: Other: SQIN

INTERVENTIONS:
Other: SQIN — Each patient will be asked to self-apply both creams (experimental vs positive control) on the right and left sides of their body (sides will be randomly assigned).
  Other Names: SQIN on one side - control cream on other side
  Arms: Experimental Cream
Other: standard moisturizing cream (Glaxal Base)
  Arms: Positive Control

SUMMARY:
In the general population, xerosis is often caused by external factors such as seasonal changes. In that case, the best way to relieve dry skin is to use a standard moisturizer. However, for those suffering of mobility problems due to age or paralysis (e.g., spinal cord injury, multiple sclerosis, Parkinson's, etc), xerosis is often severe and chronic because of the multiple causes (endogenous rather than exogenous ones) underlying such mobility impairment-related skin problems. This study is a double-blind, randomized study with positive control (active comparator) to assess the safety and efficacy of SQIN with CanSATs (Co-Activation of Natural Synergistically Acting Target-receptorS) technology on dry skin in patients suffering of paralysis.

DETAILED DESCRIPTION:
Xerosis is a medical term for dry skin. When it results in skin that is scaly and itchy, the condition is called pruritus. This occurs when natural moisture is drawn out of the skin. The skin needs moisture to protect itself. The best way to relieve dry skin normally, for those suffering of seasonal dry skin problems, is to use standard moisturizers. However, for those suffering of mobility problems due to age or paralysis (spinal cord injury, multiple sclerosis, Parkinson's, Alzheimer's, muscular dystrophy, amputation, cerebral palsy, or other comparable disorders), xerosis becomes severe and chronic because of the multiple causes (endogenous metabolic problems and dysfunctions rather than exogenous ones). SQIN with CanSATs technology is designed to act upon multiple mechanisms for enhanced protecting, moisturizing, and repairing effects. Based upon preliminary evidence, SQIN with CanSATs technology can thus elicit significantly superior effects compared with standard, commercially available moisturizers.

ELIGIBILITY:
Inclusion Criteria:

* Paralyzed due to a spinal cord injury (traumatic or non-traumatic origin)
* Chronically injured (at least 3 months post-injury)
* Paraplegic or tetraplegic
* 18-75 years of age
* Men and women
* French-speaking

Exclusion Criteria:

* Acute or subacute stage (within 1 day and 3 months post-injury)
* Had tumor(s) (malignant or non-malignant) of the skin in the last five (5) years
* Allergic or hypersensitive to any ingredient, investigational or control product
* With psychiatric or mental disorder(s)
* Children (younger than 18 year-old) or elderly (older than 75 year-old)
* Not French-speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Skin tolerance (Self-assessment of redness or itchiness problems) | 14 days
  Self-assessment of redness or itchiness problems during or after the treatment
Moisturizing level (Self-assessment (5-level score) | 14 days
  Self-assessment (5-level score) of dry skin conditions before, during and after the treatment
Elasticity level (Self-assessment (5-level score) | 14 days
  Self-assessment (5-level score) of the elasticity level of the skin before, during and after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Guertin, Ph.D., Study Director — Nordic Life Science Pipeline and Laval University
Locations (1):
- Nordic Life Science Pipeline, Québec, Quebec, Canada